CLINICAL TRIAL: NCT03301714
Title: Oral Health Education Interventions and Its Association With Behavioral Outcomes: A Clinical Trial
Brief Title: Oral Health Education Interventions Among Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Colgate Palmolive (Industry); KleinLife (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TempleU
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Quality of Life; Self Efficacy; Knowledge
Keywords: motivational interviewing; elderly; oral health
MeSH Terms: interventions — Health Education, Dental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control: Standard of Care (No Intervention): Regular dental care under the standard clinic operation
- Intervention 1: Group-based oral health education (Experimental): Group based oral health education
  Interventions: Behavioral: Oral Health Education
- Intervention 2: Individual-based oral health education (Experimental): Individual-based motivational interviewing
  Interventions: Behavioral: Oral Health Education

INTERVENTIONS:
Behavioral: Oral Health Education — Group-based oral health education vs Individual-based oral health education using motivational interviewing
  Arms: Intervention 1: Group-based oral health education; Intervention 2: Individual-based oral health education

SUMMARY:
The study aims to assess the efficacy of an oral health education group based activity versus an individual based oral health education activity in terms of changes in oral health related quality of life (OHRQoL), self-efficacy and oral health knowledge.

DETAILED DESCRIPTION:
Older adults have been described as one of the most underserved and vulnerable groups, who are at the highest risk for coronal and root caries, especially because more elderly adults are retaining their teeth. The Northeast Philadelphia KleinLife site is an important destination for the region's Jewish population comprising of at least 6500 seniors, and assisting more than 4500 seniors through food security programs. Recently, Temple University Kornberg School of Dentistry (TUKSoD) purchased the dental center at the facility to expand the services provided to these underserved population and improve their oral health. The study aims to assess the efficacy of an oral health education group based activity versus an individual based oral health education activity in terms of changes in oral health related quality of life (OHRQoL), self-efficacy and oral health knowledge. Methods: A non-probability sample of 190 senior members will be invited to participate in the trial. Potential subjects will be obtained in person through the ongoing flow of patients at TUKSoD Clinic at Kleinlife and the dental school. Seniors who consent to participate in the study will be randomly allocated to one of the 3 groups (Control: subjects will continue receiving regular dental care at the clinic, Intervention 1: subjects will continue receiving regular dental care at the clinic and be invited to participate in 2 group based education sessions during a 12 month period, and Intervention 2: subjects will continue receiving regular dental care at the clinic and be invited to participate in an individual-based education and prevention activity over a 18 month period. Randomization will be determined according to a predetermined random sequence, and neither the patient nor the research staff will be aware of the randomization outcome until after the patient has agreed to participate. The OHIP-14 will be used to assess OHRQoL, and self-efficacy scores will be the primary outcomes. Initially, we will assess the differences between the interventions and control using 2-sample t-tests. The main analysis will be based on linear mixed-effects models for repeated measures (using the OHIP 14 and self-efficacy scores as continuous outcome variables) to assess differences between intervention and control groups. Similar analyses will be conducted for secondary outcome measures Statistical significance will be set at p < .05.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 55 years old or older.
2. May be new, regular, emergency patients attending the TUKSoD clinic at Kleinlife or clinics at the Dental School or utilizing medical and social services at Kleinlife who have the intention to become patients of record at the dental clinic.
3. Must be able to speak and understand English.
4. Must be willing to provide consent to participate in the study for himself/herself.

Exclusion Criteria:

1. Subjects younger than 55 years old will be excluded from the study.
2. Subjects who do not provide consent for participation will be excluded from the study.
3. Subjects who do not speak and understand English

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MARISOL TELLEZ, PhD, Principal Investigator — Associate Professor Temple University
Locations (1):
- Temple Univerity Kornberg School of Dentistry, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention 1: Group-based Oral Health Education: Group based oral health education
  Oral Health Education: Group based oral health education vs Individual motivational interviewing
- Intervention 2:Individual-based Oral Health Education Using MI: Individual-based motivational interviewing
  Oral Health Education: Group based oral health education vs Individual motivational interviewing
Period: Overall Study
Arm/Group | Control: Standard of Care | Intervention 1: Group-based Oral Health Education | Intervention 2:Individual-based Oral Health Education Using MI
Started | 60 | 60 | 60
Completed | 50 | 54 | 53
Not Completed | 10 | 6 | 7
Not completed — Lost to Follow-up | 10 | 4 | 4
Not completed — Did not receive allocated intervention | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Control: Regular dental care under the standard clinic operation
- Intervention 1: Group based oral health education
  Oral Health Education: Group based oral health education vs Individual motivational interviewing
- Intervention 2: Individual-based motivational interviewing
  Oral Health Education: Group based oral health education vs Individual motivational interviewing
- Total: Total of all reporting groups
Arm/Group | Control | Intervention 1 | Intervention 2 | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (9.5) | 69.5 (9.1) | 69.5 (10.7) | 69.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 34 | 37 | 112
  Male | 19 | 26 | 23 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 16 | 13 | 40
  White | 41 | 41 | 39 | 121
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 2 | 6
Oral Health Related Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The oral health related quality of life scale is a 14-item measurement of individuals' perceptions of the social impact of oral conditions on their well-being. Items are rated on a 5- point Likert type scale ranging from 0 (never) to 4 (very often), regarding how frequently impact has been experienced. The total score ranges from 0 to 56; higher OHIP-14 scores indicate greater impact, hence poorer oral-health-related quality of life.
  units on a scale | 11.1 (10.5) | 14.5 (13.4) | 16.3 (13.1) | 13.9 (12.5)
Self Efficacy [Mean (Standard Deviation); unit: units on a scale] — Oral health self efficacy uses a 6 item scale and is a measurement of how confident seniors feel about their ability to perform oral hygiene tasks (1) under a lot of stress; (2) being depressed; (3) feeling anxious; (4) feeling that they were too busy; (5) being tired or; (6) being worried about other things in their life. The four response options range from 'very confident' to 'not at all confident'. The possible score range is 0 to 24,with high scores indicating high self-efficacy.
  units on a scale | 25.6 (6.5) | 23.5 (6.7) | 23.4 (7.4) | 24.2 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Oral Health Related Quality of Life (OHIP-14; Slade, 1997)
Description: The oral health related quality of life scale is a 14-item measurement of individuals' perceptions of the social impact of oral conditions on their well-being. This scale evaluates the consequences of oral conditions across dimensions of functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Items are rated on a 5- point Likert type scale ranging from 0 (never) to 4 (very often), regarding how frequently impact has been experienced. The total score ranges from 0 to 56; higher OHIP-14 scores indicate greater impact, hence poorer oral-health-related quality of life.
Time Frame: change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention 1 | Intervention 2
Number analyzed (Participants) | 60 | 60 | 60
score on a scale | 16.8 (11.4) | 12.4 (11.2) | 10.5 (10.5)
Statistical Analysis 1: Comparison: Control vs Intervention 1 vs Intervention 2; Test type: Equivalence — equivalence analysis; p = .000, Regression, Linear — baseline demographics, correlated errors due to repeated measures, and bias due to lost to follow-up were accounted for via Generalized Estimating Equation (statistical threshold <0.01); Mean Difference (Final Values) = 7.62 — Mean change difference in oral health related quality of life among control, intervention 1: group-based oral health education and intervention 2: individual-based oral health education using motivational interviewing

2. Primary Outcome: Change in Oral Health Self Efficacy (Modified Version of Finlayson, 2007).
Description: Oral health self efficacy uses a 6 item scale and is a measurement of how confident seniors feel about their ability to perform oral hygiene tasks (1) under a lot of stress; (2) being depressed; (3) feeling anxious; (4) feeling that they were too busy; (5) being tired or; (6) being worried about other things in their life. The four response options range from 'very confident' to 'not at all confident'. The possible score range is 0 to 24,with high scores indicating high self-efficacy.
Time Frame: change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention 1 | Intervention 2
Number analyzed (Participants) | 60 | 60 | 60
score on a scale | 23.5 (6.6) | 24.5 (7.5) | 27.6 (5.9)

3. Secondary Outcome: Change in Oral Health Knowledge (Khanagar, 2014)
Description: Oral health knowledge measurement of the seniors pre and post intervention will be conducted using a list of 15 knowledge statements to which subjects had to report agreement wit the statement (yes), disagreement (no) or don't know. The frequency numbers provided in the results table correspond to correct responses for each individual item.
Time Frame: change from baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control: Standard of Care | Intervention 1: Group-based Oral Health Education | Intervention 2: Individual-based Oral Health Education
Number analyzed (Participants) | 60 | 60 | 60
Participants
  When gums bleed during brushing.... | 9 | 11 | 12
  health of mouth directly related to body.. | 48 | 43 | 46
  You can chew just as well with dentures as with | 15 | 19 | 16
  Older adults with dry mouth get more cavities | 29 | 18 | 18
  The most common cause of dry mouth is medication | 31 | 33 | 27
  It is normal for people to have pain and sores in | 7 | 10 | 8
  Individuals who do not cooperate for daily mouth c | 5 | 7 | 5
  Name Box Insert Function Dental check-ups are as i | 52 | 54 | 52
  People can lose their teeth if they remain dirty | 48 | 45 | 48
  As people get old they naturally lose their teeth | 19 | 23 | 23
  Dentures that don't fit well can cause oral cancer | 12 | 10 | 16
  Dentures should be removed for few hours every day | 26 | 26 | 27
  People with no teeth need to be seen by dentist | 41 | 35 | 39
  Mouth rinsing is a good alternative to daily tooth | 12 | 21 | 20
  Older adults with teeth need to use fluorides | 35 | 38 | 31

ADVERSE EVENTS:
Time Frame: No adverse event data were collected.
Description: No adverse event data were collected.Nature of intervention tested would not generate mortality outcomes.
Arm/Group | Control | Intervention 1 | Intervention 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT03301714/Prot_SAP_000.pdf